CLINICAL TRIAL: NCT06548243
Title: Act With Nature (AWN): Promoting Well-being and Pro-environmental Behaviour Among Working-age Adults During the Era of Environmental Crises
Brief Title: Act With Nature: Promoting Planetary Well-being
Acronym: AWN
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: JAMK University Of Applied Sciences (Other)
Collaborators: Tampere University (Other); University of Surrey (Other)
Responsible Party: Principal Investigator, Katriina Hyvonen, Senior Researcher, PhD, Adj. Prof., JAMK University Of Applied Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: JAMKUAS_AWN
Record Dates: First submitted 2024-08-07; First posted 2024-08-12 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2024-08

CONDITIONS: Well-Being, Psychological
Keywords: Pro-environmental behaviour; Nature-based programme; Nature connectedness; Environmental emotions
MeSH Terms: conditions — Psychological Well-Being | interventions — alpha 1-Antichymotrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Act with Nature Programme (Experimental): A nature-based programme to promote well-being and pro-environmental behaviour. The programme is facilitated by a trained health care professional.
  Interventions: Behavioral: Act with Nature Programme
- Control group (No Intervention): The participants in the control group continue life as usual.

INTERVENTIONS:
Behavioral: Act with Nature Programme — The participants in the intervention group are offered a 12-week nature-based programme, which includes independent exercises and information on an online learning environment, as well as online or in-person group meetings.
  Arms: Act with Nature Programme

SUMMARY:
The research investigates the effects of nature-based programme (Act with Nature; AWN) in promoting psychological well-being and pro-environmental behaviour among working age participants in Finland. Our research deepens understanding of how coping with environment-related emotions and nature connectedness are connected to human wellbeing and pro-environmental behaviour. The psychological wellbeing and pro-environmental behaviour are investigated with self-report measures and analysed with quantitative and qualitative methods. The project will provide a new programme (AWN) for combining individual well-being and behaviour change. The results can provide a theoretical framework and working model for health professionals to intervene and support people in adapting to environmental crises and coping with stress.

DETAILED DESCRIPTION:
An intervention study with a randomised control trial design will be conducted among a sample of 158 working age participants in various locations in Finland. After receiving information about the research and signing the study consent, participants are randomly allocated to intervention and control groups. The participants in the intervention group will be offered a 12-week, nature-based, Act with Nature (AWN) programme. The programme will be carried out online with individual coaching and independent tasks for each week. Participants share experiences during workshops that are facilitated in nature environment, either in-person or online.

Throughout the AWN programme, nature-based exercises are facilitated in which participants are encouraged to recognise the significance of physical environment and social support in coping with environment-related emotions, nature connectedness and wellbeing. AWN programme is facilitated by a trained health care professional.

The AWN has three separate stages (4 weeks each): Stage 1: nature connectedness, environmental self-regulation and confidence in the group; Stage 2: environmental-related emotions, psychological flexibility and coping strategies; Stage 3: experimenting with change alternatives and affirming positive change in environmental behaviour.

Participants respond to online surveys at five measurement points: a pre-measurement at the start of the programme, two measurements during the programme (at 4 and 8 weeks of the programme), a post-measurement at the end of the programme, and a follow-up measurement three months after the end of the programme. The participants in the intervention group (nature-based AWN programme) are compared to the participants in the control group who continue life as usual and only respond to online surveys at three measurement points (pre-, post- and follow-up measurements). Coping with environment-related emotions, comprehensive nature experience, nature connectedness, environmental emotions and personal environmental goals are investigated as mediators to explain changes in well-being and pro-environmental behaviour.

This research is funded by the Research Council of Finland (Project Numbers: 350971 and 350964).

ELIGIBILITY:
Inclusion Criteria:

* Working age adults
* Able to communicate adequately in Finnish in order to participate
* Willingness to commit to a 12-week intervention programme

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 158 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Emotional wellbeing | 6 months
  Health related quality of life (RAND): emotional wellbeing dimension, the scores range from 1 to 6 and some items are recoded. Higher total score refers to better emotional wellbeing.
Mental wellbeing | 6 months
  Short Warwick-Edinburgh Mental Well-being Scale (SWEMWBS), the scores range from 1 to 5, a higher scores refers to better mental wellbeing.
Pro-environmental behaviour | 6 months
  Self-report scale of the frequency of pro-environmental actions. Items refering to pro-environmental actions during one month are responded on a scale ranging from 1 to 5. Items refering to pro-environmental actions during the past year are responded on a scale 1 (yes) and 2 (no). Some items are recoded and all items include an option for "doesn't apply to me". A higher total score refers to more self-reported pro-environmental behaviour.

SECONDARY OUTCOMES:
Behavioural Willingness | 6 months
  Willingness to act pro-environmentally, the scores range from 1 to 4. A higher score refers to more willingness to act pro-environmentally.
Affect regulation | 6 months
  Measure of Affect Regulation Styles (MARS), the scores range from 1 to 6 and all items include an option for "doesn't apply to me". A higher score refers to a higher efficiency in affect regulation styles.

CONTACTS AND LOCATIONS:
Overall Officials: Katriina Hyvönen, PhD, Principal Investigator — JAMK University Of Applied Sciences
Locations (2):
- Finland (2):
  - Institute of Rehabilitation, JAMK University of Applied Sciences, Jyväskylä
  - Tampere University, Tampere

IPD SHARING:
Plan to Share IPD: Yes
Data from surveys will be anonymised after the research and will be archived to the research data storage service (IDA). Anonymised data will open for reuse after the research finishes in 2026. The reuse of interview data will be restricted to suitable parts.
Supporting Information: Study Protocol

REFERENCES:
- [Background] Korpela, K., Hyvönen, K., Ratcliffe, E., Salonen, K., & Paakkolanvaara, J.-V. (2023, Jan 30). Act with Nature (AWN): Promoting well-being and pro-environmental behaviour among working-age adults during the era of environmental crises. https://doi.org/10.17605/OSF.IO/69QVW
- See also: Project website — http://www.jamk.fi/en/research-and-development/rdi-projects/act-with-nature-awn-promoting-well-being-and-pro-environmental-behaviour-among-working-age-adults
- See also: Project website — http://research.tuni.fi/enviwell/projects/
- See also: OSF Preregistration of the research — https://doi.org/10.17605/OSF.IO/69QVW